CLINICAL TRIAL: NCT01358292
Title: Semi-extended Position vs. 90 Degrees of Flexion for Intramedullary Nailing of the Tibia: a Randomized Clinical Trial
Brief Title: Efficacy Study of Surgical Technique in Intramedullary Tibia Nailing, Using Trigen META Tibia Nails
Acronym: TrigenMETA
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Smith & Nephew Orthopaedics AG (Industry)
Responsible Party: Sponsor
Organization: Smith & Nephew, Inc. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: R11021-1
Record Dates: First submitted 2011-01-14; First posted 2011-05-23 (Estimated); Last update posted 2016-06-17 (Estimated); Status verified 2015-11

CONDITIONS: Tibial Fractures
Keywords: Intramedullary tibia nailing; Anterior Knee Pain; Nail positioning
MeSH Terms: conditions — Tibial Fractures

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Semi-extended surgical technique (Experimental): The experimental technique for implanting an intramedullary tibia nail is with the knee in 10-20 degrees of flexion.
  Interventions: Procedure: Semi-extended Surgical Technique
- Standard Surgical Technique (Active Comparator): The standard surgical technique in intramedullary tibia nailing is with the knee in almost 90 degrees of flexion.
  Interventions: Procedure: Standard Surgical Technique

INTERVENTIONS:
Procedure: Semi-extended Surgical Technique — Surgical technique with the knee in 10-20 degrees of flexion, to implant the intramedullary tibia nail.
  Other Names: Trigen META Intramedullray Tibia Nail
  Arms: Semi-extended surgical technique
Procedure: Standard Surgical Technique — Th e Standard surgical techique is implanting the tibia nail with the knee in 90 degrees of flexion.
  Other Names: Trigen META intramedullary tibia nailing
  Arms: Standard Surgical Technique

SUMMARY:
Multicentre Prospective Randomized Clinical Trial, to evaluate patients after surgery for extra-articular tibial fractures treated with Smith& Nephew's Trigen META intramedullary nailing system; comparing two surgical techniques: Group A=standard technique(90º of knee flexion) and Group B=with the semi-extended surgical technique. (2*100 patients)

Research Objectives:

The primary research objectives are to evaluate:

i) anterior knee pain and ii) the nail position and overall fracture alignment

Outcome Measures:

1. Nail positioning by means of intra-operative fluoroscopy and post operative x-rays.
2. Anterior Knee pain by means of VAS-scores, a Kneeling test and Subjective outcomes by means of Patient questionnaires
3. Knee-related adverse events
4. Overall fracture alignment

DETAILED DESCRIPTION:
After surgery with standard intramedullary nailing technique in tibia fractures, 40-80% of the patients still complain of anterior knee pain postoperative. The expected advantages of the semi-extended nailing technique is less anterior knee pain and less malunion of the fracture.

Using the semi-extended nailing technique also might give the advantage of better position of the nail by a more concentric reaming of the tibia, due to less tension on the patella tendon during reaming process.

ELIGIBILITY:
Inclusion Criteria:

* Patient has sustained a closed (Tscherne Classification) or open tibial fracture (Gustillo-Anderson Classification) that is amendable for operative fixation with an intramedullary nail.
* Patient has an isolated tibia and fibula fracture
* Skeletally mature
* Patients aged between/including 18 to 70 years
* Patient has given formal consent to be involved in the trial and has completed the study consent form
* Patient is likely to comply with study follow-up requirements

Exclusion Criteria:

* Pathologic fractures
* Other fractures involving the same lower extremity
* Soft tissue injuries/problems that would prevent the surgeon from using both of the surgical techniques to insert an intramedullary nail
* Patient having pre-existing knee joint disease causing anterior knee pain
* Patient likely to have problems with follow-up
* Patient unwilling to give informed consent to be included in the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 95 (Actual)
Dates: Start 2011-02; Primary Completion 2015-09 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Anterior Knee Pain | 4, 6 and 12 months post-operative
  Anterior Knee pain will be measured through a Kneeling test (time a patient is able to rest on his operated knee)

SECONDARY OUTCOMES:
Nail positioning | Operation (day 1)
  Measure by means of fluoroscopy and standard x-rays during the surgery, the position of both the guide wire and the intramedullary nail.

CONTACTS AND LOCATIONS:
Overall Officials: Alan Johnstone, Professor, Principal Investigator — Aberdeen Royal Infirmary; Pedro Caba, Dr., Study Chair — Hospital de 12 Octubre, Madrid; Markus Graf, Dr., Study Chair — Medizinisches Zentrum StädteRegion Aachen; Ismael Escriba, Dr., Study Chair — Hospital La Fe de Valencia; Daren Forward, MA, FRCS, DM, Study Chair — Nottingham University Hospital
Locations (5):
- Medizinisches Zentrum StädteRegion Aachen, Würselen, Germany
- Spain (2):
  - Hoisptal de 12 Octubre, Madrid
  - Hospital La Fe, Valencia
- United Kingdom (2):
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Nottingham University Hospitals, Nottingham

IPD SHARING:
Plan to Share IPD: No